CLINICAL TRIAL: NCT06922136
Title: A Prospective, Randomized, Controlled, 2-arms, Double-blind, Multicentre Clinical Investigation to Evaluate the Performance and Safety of Hyalo Gyn® Gel Compared to Placebo in the Management of Vulvovaginal Atrophy in Postmenopausal Breast Cancer Survivors
Brief Title: Evaluation of the Performance and Safety of Hyalo Gyn® Gel Compared to Placebo in Postmenopausal Breast Cancer Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QQ53-21-01
Record Dates: First submitted 2025-03-17; First posted 2025-04-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Vulvo Vaginal Atrophy

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, 2-arms, placebo-controlled, double-blind, multicentre clinical investigation
Who Masked: Participant, Investigator
Masking Description: The double-blind design for this investigation was made possible by means of the realisation of a placebo that is indistinguishable from the active Hyalo Gyn® gel in terms of shape, colour, consistency, small and mode of application, in order that neither the Investigator nor the study staff, nor the patient will be aware of the assigned treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Hyalo Gyn® Gel (Experimental): Hyalo Gyn® vaginal gel is formulated with Hydeal-D®, a proprietary HA derivative component
  Interventions: Device: Hyalo Gyn Vaginal Gel
- Group B: Placebo (Placebo Comparator): Matched plecebo A
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Hyalo Gyn Vaginal Gel — Hyalo Gyn® is uniquely formulated with Hydeal-D®, a proprietary HA derivative component manufactured by Fidia Farmaceutici S.p.A.
  Arms: Group A: Hyalo Gyn® Gel
Other: Placebo — Placebo
  Arms: Group B: Placebo

SUMMARY:
Eligible patients will be randomized to treatment with Hyalo Gyn® gel or placebo, at the dose regimen of 1 application deeply in the vagina every 3 days (i.e. an application is followed by 2 days without application), up to a total of 12 consecutive weeks.

After 12 weeks (i.e. at Visit 3), the following rules will apply for the second 12- week phase of the study:

* In case of resolution of the symptom (the dryness single score is equal to zero), the patient will suspend treatment and will undergo follow-up visits;
* In case of the single score is reduced but still greater than zero: the subject will receive Hyalo Gyn® open-label.
* In case the dryness gets worse the subject can choose whether receive Hyalo Gyn® gel open-label or undergo the follow-up visits. Patients will be allowed to use only water-based lubricants, not containing HA, hormones, or isoflavones, if necessary, only when engaging in sexual activity and specifying the reason for its use (multiple choice answer). The number of lubricant applications, as well as the frequency of the sexual activity, will be recorded weekly in the diary by the patient.

DETAILED DESCRIPTION:
This will be a prospective, randomized, controlled, 2-arms, placebo-controlled, double-blind, multicentre clinical investigation. Patients with good compliance and who are voluntary to sign the informed consent will be enrolled in a period time of approximately 6 months. The screened and eligible patients will be randomly assigned in one of the two groups: Group A will receive Hyalo Gyn® and Group B will receive Placebo. Neither the Investigator nor the Patient will be aware of the assigned treatment.

Subjects of both groups will start the treatment with 1 application of Hyalo Gyn® gel or placebo gel, deeply in the vagina every 3 days (i.e. an application is followed by 2 days without application) up to a total of 12 consecutive weeks.

After 12 weeks (i.e. at Visit 3), according to the status of dryness symptom, measured with the VRS dryness score from baseline to 12 weeks, patients will undergo different procedures for the second phase of the study as reported in the brief summary.

Visits at the investigational site will be performed at screening/baseline (V0, Week 0) and every 4 weeks, alternated to telephone contacts by the clinician (V1, Week 4; T1, Week 6; V2, Week 8; T2, Week 10; V3, Week 12) up to the end of the first 12-week phase of the study. Two phone follow-up visits will be performed at Week 16 (T3) and Week 20 (T4), followed by a visit at the investigational site at the end of the second 12-week phase of the study (V4, Week 24). Visit 4 (Week 24) will represent the end of study visit. In case of premature withdrawal from the investigation for whatever reason an "Early termination Visit" will be performed, which will include all assessments foreseen for the final visit (Visit 4, Week 24 ± 5 days).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to beginning specific protocol procedures;
2. Women between 25 and 80 years of age (inclusive);
3. Women with intention or willingness to have sex;
4. Patients with a history of breast cancer who had completed primary cancer treatment (surgery, non-endocrine chemotherapy, or radiation therapy) 3-60 months prior to enrolment;
5. Patient receiving endocrine therapy (an AI or tamoxifen or a GnRH analogue) as a breast cancer treatment in the adjuvant setting for a minimum of 3 months. The therapy program must cover the entire duration of the study (24 weeks);
6. Life expectancy of at least 12 months;
7. Postmenopausal status defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum follicle stimulating hormone (FSH) levels > 40 mIU/ml or 6 weeks' postsurgical bilateral oophorectomy with or without hysterectomy;
8. Vulvovaginal dryness assessed as moderate to severe. A moderate and severe symptom (i.e. a score of 2 = moderate or 3 = severe) will be considered if the symptoms are present and could be bothersome and could interfere with the normal patient activity;
9. Vaginal Health Index ≤15;
10. Vaginal pH ≥5;
11. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1;
12. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures;
13. Patients legally able to give written informed consent to the trial (signed and dated by the participant) and able to understand study procedures and protocol requirements.

Exclusion Criteria:

1. Stage IIIB-IV breast cancer;
2. Treatment with any other current anti-tumoral therapy besides an AI or tamoxifen or a GnRH analogue;
3. Prior history of other malignancy other to breast cancer within 5 years of study entry, with the exception of non-melanoma skin cancer or carcinoma in-situ of the uterine cervix adequately treated;
4. Postmenopausal uterine bleeding and/or vaginal bleeding of unknown aetiology;
5. Patients with endometrial thickness equal to or greater than 4 mm for patientson AI or GnRH analogue, or equal to or greater than 9 mm for patients on tamoxifen, measured by transvaginal ultrasound;
6. Patients who have received any type of vulvovaginal treatment in the 15 days prior to the start of the study;
7. Patients that present clinical signs of vaginal infections such as trichomonas, candida, and bacterial vaginosis (BV), confirmed with a vaginal swab;
8. Patients with a history of vulvovaginal contact allergy or with a diagnosis of vulvovaginal lichen;
9. Positive history of hypersensitivity to hyaluronic acid (HA) or to any component of the medical device;
10. Use of any hormone, or any products with phytoestrogenic activity (for instance resveratrol, flax seeds, hops, isoflavones as red clover and soy) for the treatment of menopausal symptoms in the previous month (cimicifuga extract and pollen are allowed);
11. Known human immunodeficiency virus infection;
12. Other severe acute or chronic medical condition, or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with investigation participation or product administration and investigation's procedures, or which, in the judgment of the investigator, would make the patient inappropriate for entry into this investigation;
13. Previous investigational treatment for any condition or participation in any clinical trial in the previous month before inclusion date

Ages: 25 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-01-30 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the performance of Hyalo Gyn® vaginal gel in the improvement of patient's perception of vulvovaginal dryness associated with vulvovaginal atrophy, after 12 weeks of treatment, compared to placebo. | after 12 weeks of treatment
  The primary performance endpoint of the investigation will be the change in the vulvovaginal dryness associated with vulvovaginal atrophy, evaluated as the proportion of subjects having a reduction ≥2 points in the Verbal Rating Scale (VRS) dryness score from baseline to 12 weeks of treatment with Hyalo Gyn® gel compared to placebo. The vulvovaginal symptom associated with vulvovaginal atrophy (dryness) will be reported on a four-point scale (0 = absent, 1 = mild, 2 = moderate, 3= severe).

SECONDARY OUTCOMES:
Change from baseline in patient's perception of dryness, irritation/itching, soreness, dysuria, and dyspareunia vulvovaginal symptoms single scores associated with vulvovaginal atrophy | After 4, 6, 8, 10, and 12 weeks of treatment from baseline (V0)
  Change from baseline in the vulvovaginal symptoms associated with vulvovaginal atrophy, evaluated by measuring the VRS single score at baseline and at 4, 6, 8, 10, and 12 weeks of treatment with Hyalo Gyn® gel compared to placebo. Each vulvovaginal symptom associated with vulvovaginal atrophy (dryness, irritation/itching, soreness, dysuria, dyspareunia) will be reported on a four-point scale (0 = absent, 1= mild, 2 = moderate, 3 = severe);
Change from baseline in patient's perception of vulvovaginal symptoms global score associated with vulvovaginal atrophy; | After 4, 6, 8, 10, and 12 weeks of treatment from baseline (V0)
  Change from baseline in the vulvovaginal symptoms associated with vulvovaginal atrophy, evaluated by measuring the VRS global score at baseline and at 4, 6, 8, 10, and 12 weeks of treatment with Hyalo Gyn® gel compared to placebo. Each vulvovaginal symptom associated with vulvovaginal atrophy (dryness, irritation/itching, soreness, dysuria, dyspareunia) will be reported on a four-point scale and the sum of every single score will be calculated (0 = absent,
  1= mild, 2 = moderate, 3 = severe);
Change from baseline of sexual function through Female Sexual Function Index (FSFI) questionnaire | After 4, 8 and 12 weeks of treatment from baseline (V0)
  Change from baseline in the sexual function, evaluated with the questionnaire FSFI at 4, 8, and 12 weeks of treatment with Hyalo Gyn® gel compared to placebo. The FSFI questionnaire consists of 19 items (six subscales: desire, arousal, lubrication, orgasm, satisfaction, and pain). Total scores range from 2 to 36, with higher scores reflecting better sexual function (cut-off value = 26.5).
Change from baseline of sexual function through Female Sexual Distress Scale-Revised (FSDS-R) questionnaire | After 4, 8 and 12 weeks of treatment from baseline (V0)
  Change from baseline in the sexual distress, evaluated with the FSDS-R at 4, 8, and 12 weeks of treatment with Hyalo Gyn® gel compared to placebo. The FSDS-R questionnaire consists of 13 items and items are scored on a five-point rating scale (0 = never; 1 = rarely; 2 = occasionally; 3 = frequently; 4 = always). Total score ranges from 0 to 52, with higher scores indicating greater sexual distress (cut-off value = 11);
Change from baseline of Vaginal Health Index (VHI); | After 4, 8 and 12 weeks of treatment from baseline (V0),
  Change from baseline in vaginal signs associated with vulvovaginal atrophy, evaluated by measuring the average score of VHI at baseline and at 4, 8, and 12 weeks of treatment with Hyalo Gyn® gel compared to placebo. The VHI will be calculated assigning a score between 1 to 5 for vaginal moisture, vaginal fluid volume, vaginal elasticity, vaginal pH, and vaginal epithelial integrity on a scale of 1 to 5. The assigned score will vary from 5 to 25. The lower the score, the greater the atrophy (cut-off value = 15).
Change from baseline of the objective genitourinary atrophy signs (Vaginal Maturation Index (VMI, only after 12 weeks); | After 4, 8 and 12 weeks of treatment from baseline (V0
  Change from baseline of the objective genitourinary atrophy sign VMI, evaluated at baseline and at 12 weeks of treatment with Hyalo Gyn® gel compared to placebo. VMI quantifies the percentages of parabasal, intermediate, and superficial cells by using the formula: VMI = [1(% superficial cells)] + [0.6(% intermediate cells)] + [0.2(% parabasal cells)] (0%-49%, low stimulation of the vaginal epithelium; 50%-64%, moderate stimulation of the vaginal epithelium; 65%-100%, high stimulation of the vaginal epithelium).
Change from baseline of the objective genitourinary atrophy sign, vaginal pH | After 4, 6, 8, 10, and 12 weeks of treatment from baseline (V0)
  Change from baseline of the objective genitourinary atrophy sign vaginal pH, evaluated by measuring values of vaginal pH at baseline and at 4, 8, and 12 weeks of treatment with Hyalo Gyn® gel compared to placebo. The pH values will be grouped in a 4-point scale and scored respectively: pH < 5 (0), 5-5.49 (1), 5.5- 6.49 (2), and more than 6.49 (3)
Evaluation of Patient's global assessment (PTGA) of overall satisfaction | After 4, 8, and 12 weeks of treatment from baseline (V0)
  PTGA of overall satisfaction, evaluated at 4, 8, and after 12 weeks of treatment with Hyalo Gyn® gel compared to placebo. The patient will be requested to score the overall satisfaction of the treatment on a four-grade scale: 0 = dissatisfied or very dissatisfied, 1 = moderately satisfied or satisfied, 2 = very satisfied, and 3 = greatly satisfied
Evaluation of the safety and tolerability of Hyalo Gyn® vaginal gel compared to placebo during the entire course of the study | After 4, 6, 8, 10, and 12 weeks of treatment from baseline (V0)
  Safety of the treatment, evaluated at 4, 6, 8, 10, and 12 weeks of treatment by tracking the number of patient withdrawals and collecting the local and general adverse events that occur during the study

CONTACTS AND LOCATIONS:
Locations (7):
- Italy (7):
  - Policlinico SantOrsola Malpighi, Bologna, BO
  - AOUC Azienda Ospedaliero-Universitaria Careggi, Florence, FI
  - Azienda Ospedaliera-Universitaria UOC Clinica Ginecologica e Ostetrica dell'Università, Padua, PD
  - Fondazione IRCCS Policlinico San Matteo, Pavia, PV
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, RM
  - AO Ordine Mauriziano di Torino, Ospedale Umberto I, Torino, TO
  - Istituto Europeo di Oncologia, Milan

IPD SHARING:
Plan to Share IPD: No